CLINICAL TRIAL: NCT00863759
Title: Wavefront Analysis and Contrast Sensitivity After Cataract Surgery With Akreos AO Intraocular Lens Implantation: Clinical Comparative Study
Brief Title: Wavefront Analysis and Contrast Sensitivity After Cataract Surgery With Akreos Advanced Optics Intraocular Lens Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Marcony Santhiago, MD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 656/06
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2009-03

CONDITIONS: Lens Implantation, Intraocular
Keywords: intra-ocular lenses; comparative study; Ocular aberrations; Contrast Sensitivity
MeSH Terms: interventions — Lens Implantation, Intraocular

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients will receive an aspheric intraocular lenses (IOL) Akreos AO in the right eye and an spheric IOL Akreos Fit in the left eye, during cataract surgery.
  Interventions: Procedure: implantation of intraocular lens (IOL)
- 2 (Active Comparator): Patients will receive an spheric intraocular lens (IOL) Akreos Fit in the right eye and an aspheric IOL Akreos AO in the left eye, during cataract surgery.
  Interventions: Procedure: implantation of intraocular lens (IOL)

INTERVENTIONS:
Procedure: implantation of intraocular lens (IOL) — implantation of intraocular lens during cataract surgery.
  Arm 1: implantation of aspheric IOL Akreos AO in right eye and an spheric IOL Akreos Fit in left eye.
  Arm 2: implantation of aspheric IOL Akreos AO in left eye and an spheric IOL Akreos Fit in right eye.
  Other Names: Implantation of aspheric Akreos AO intraocular lenses (IOL); Implantation of spheric Akreos Fit intraocular lenses (IOL)

SUMMARY:
Purpose: To determine whether implantation of an intraocular lens (IOL) with a modified anterior and posterior aspherical surface (Akreos AO, Bausch & Lomb,Inc) results in reduced ocular aberrations (spherical aberration) and in improved contrast sensitivity after cataract surgery.

Study hypothesis: the implantation of an intraocular lens (IOL) with a modified anterior and posterior aspherical surface (Akreos AO, Bausch & Lomb,Inc) results in reduced ocular aberrations (spherical aberration) and improved contrast sensitivity after cataract surgery.

Setting: Department of ophthalmology, Hospital das Clínicas, University of São Paulo, São Paulo, Brazil.

Overall Study design: This will be an intraindividual randomized double-blinded prospective study. Patients will be randomized to receive an aspheric IOL Akreos AO in one eye (25 eyes; Bausch & Lomb, Inc), and an spheric IOL Akreos Fit (25 eyes; Bausch & Lomb, Inc.) in the fellow eye. Ocular aberrations with a 5.0 mm and 6.0 mm pupil will be measured with a dynamic retinoscopy aberrometer after 1 and 3 months. Uncorrected and best-corrected visual acuity, out-focus performance and contrast sensitivity under mesopic and photopic conditions will be also measured. All patients will be followed for 3 months.

DETAILED DESCRIPTION:
Patients with bilateral visually significant cataract with corneal astigmatism lower than 2.0D (diopters) will be eligible for inclusion in the study. Exclusion criteria will be any ocular diseases, such as corneal opacities or irregularity, dry eye, amblyopia, anisometropia, glaucoma, retinal abnormalities, surgical complications, IOL tilt, IOL decentration greater than 0.4 mm (estimated by retroillumination), or incomplete follow-up.

Patients will be examined before surgery and at 1, 7, 30, 90 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bilateral visually significant cataract with corneal astigmatism lower than 2.0D (diopters)

Exclusion Criteria:

* Ocular diseases, such as corneal opacities or irregularity, dry eye amblyopia, anisometropia, glaucoma, retinal abnormalities
* Surgical complications
* Intraocular lens (IOL) tilt, IOL decentration greater than 0.4 mm (estimated by retroillumination)
* Incomplete follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Ocular aberrations with a 5.0 mm and 6.0 mm pupil measured with a dynamic retinoscopy aberrometer | At 30 and 90 days postoperatively

SECONDARY OUTCOMES:
Days contrast sensitivity under photopic and mesopic conditions | at 90 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Marcony R Santhiago, MD, Principal Investigator — University of Sao Paulo (ophthalmology department of Hospital das Clinicas)
Locations (1):
- : Department of ophthalmology, Hospital das Clinicas, University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Montes-Mico R, Ferrer-Blasco T, Cervino A. Analysis of the possible benefits of aspheric intraocular lenses: review of the literature. J Cataract Refract Surg. 2009 Jan;35(1):172-81. doi: 10.1016/j.jcrs.2008.09.017. PMID 19101441
- [Background] Tzelikis PF, Akaishi L, Trindade FC, Boteon JE. Spherical aberration and contrast sensitivity in eyes implanted with aspheric and spherical intraocular lenses: a comparative study. Am J Ophthalmol. 2008 May;145(5):827-33. doi: 10.1016/j.ajo.2007.12.023. Epub 2008 Mar 4. PMID 18291345
- [Background] Kasper T, Buhren J, Kohnen T. Intraindividual comparison of higher-order aberrations after implantation of aspherical and spherical intraocular lenses as a function of pupil diameter. J Cataract Refract Surg. 2006 Jan;32(1):78-84. doi: 10.1016/j.jcrs.2005.11.018. PMID 16516783
- [Background] Dietze HH, Cox MJ. Limitations of correcting spherical aberration with aspheric intraocular lenses. J Refract Surg. 2005 Sep-Oct;21(5):S541-6. doi: 10.3928/1081-597X-20050901-24. PMID 16209458